CLINICAL TRIAL: NCT01352234
Title: Evaluation of Dose-response Effect of Acetylsalicylic Acid on Placental Development, Preterm Birth, Fetal Growth and Hypertension in Pregnancy in Women With Previous History of Preeclampsia
Brief Title: Comparison of Doses of Acetylsalicylic Acid in Women With Previous History of Preeclampsia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C10-11-108
Record Dates: First submitted 2011-04-01; First posted 2011-05-11 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Pre-Eclampsia; Fetal Growth Retardation; Premature Birth; Placental Insufficiency
MeSH Terms: conditions — Pre-Eclampsia; Fetal Growth Retardation; Premature Birth; Placental Insufficiency | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Acetylsalicylic Acid 160mg administered at bedtime
  Interventions: Drug: Acetylsalicylic Acid 160 mg
- Group B (Active Comparator): Acetylsalicylic Acid 80mg administered at bedtime
  Interventions: Drug: Acetylsalicylic Acid 80 mg

INTERVENTIONS:
Drug: Acetylsalicylic Acid 160 mg — Capsule containing Acetylsalicylic Acid 160mg pill with lactose
  Other Names: Asaphen; Aspirin; ASA
  Arms: Group A
Drug: Acetylsalicylic Acid 80 mg — Capsule containing Acetylsalicylic Acid 80mg pill with lactose
  Other Names: Asaphen; Aspirin; ASA
  Arms: Group B

SUMMARY:
Placental insufficiency is the source of preeclampsia (PE) and intrauterine growth retardation (IUGR). Current data demonstrate a significant beneficial effect of prophylactic use of aspirin on the recurrence of placental insufficiency and its complications, mainly preeclampsia, when started early in pregnancy. However, there is a significant heterogeneity in medical practice in Canada and around the world in terms of the dose of aspirin used.

The objectives of this study are: 1) Evaluate whether a dose of 160 mg of aspirin is associated with greater improvement in placental function assessed by biochemistry (sFlt-1 and endoglin) and ultrasound (uterine artery Doppler) than a dose of 80 mg in women with a history of PE, 2) Assess whether the change is dependent on platelet aggregation measured by a test used in several Canadian centers (PFA-100).

DETAILED DESCRIPTION:
Many studies suggest that aspirin (acetylsalicylic acid) at low dose significantly reduces the incidence of preeclampsia. More recent data have shown that, when administered before 16 weeks of pregnancy, aspirin can prevent over 50% of preeclampsia, severe preeclampsia, and IUGR but also a significant proportion of the rate of preterm births. Current data also demonstrate a beneficial effect of prophylactic use of aspirin when started early in pregnancy in populations composed of high-risk patients with a history of preeclampsia and / or other pregnancy complications related to poor placental function.

Beside, many clinicians are already using aspirin in the context of a proven benefit. However, the usual dose prescribed in Canada today is 80 mg while the most favorable studies have used a slightly higher dose of aspirin (100 mg).

Moreover, it has been demonstrated that the time of day during which aspirin was administered was also a very important factor regarding the effect on blood pressure and adverse outcomes of the majority of pregnancy. Yet the majority of studies in this context have not specified the time of day at which aspirin was or had been taken, possibly underestimating the effect thereof.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 10 0 / 7 and 13 6 / 7 weeks
* History of preeclampsia (as defined by The Society of Obstetricians and Gynaecologists of Canada) confirmed by medical records

Exclusion Criteria:

* Negative Fetal Heart
* Multiple pregnancy
* Anaphylactic allergy to lactose
* Kown coagulopathy (antithrombin III deficiency, factor V Leiden, antiphospholipid syndrome, the prothrombin mutation, deficiency of protein S or protein C)
* Use of heparin or other anticoagulants.
* Contraindications to aspirin
* Severe fetal abnormality (cystic hygroma, nuchal translucency> 95th percentile, anencephaly, etc.)
* History or active peptic ulcer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2011-09; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Placental function | 22nd week of gestation
  We chose a continuous intermediate variable focused on the aetiology, the placental function, assessed by Doppler ultrasound: the average pulsatility index of uterine arteries (UTAP - primary outcome) at 22 weeks of gestation

SECONDARY OUTCOMES:
Rates of pregnancy complications related to placental insufficiency (preeclampsia, IUGR, premature birth) | At delivery
  The effectiveness of treatment on the rate of preterm delivery, hypertensive disorders of pregnancy and IUGR will also be measured by reviewing medical records. All cases with a diagnosis of preterm labor, gestational hypertension or IUGR <10th percentile will be reviewed by a specialist in maternal fetal medicine at blindness for allocation.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Bujold, MD, MSc, Principal Investigator — CHU de Quebec-Universite Laval
Locations (1):
- Centre Hospitalier Universitaire de Québec (CHUQ)/Pavillon CHUL, Québec, Canada

IPD SHARING:
Plan to Share IPD: Undecided